CLINICAL TRIAL: NCT02832245
Title: Computerized Registry of Patients With Venous Thromboembolism (RIETE)
Acronym: RIETE
Status: Recruiting | Type: Observational
Sponsor: Manuel Monreal (Other)
Responsible Party: Sponsor-Investigator, Manuel Monreal, Professor of Internal Medicine, Foundation for the study of VTE diseases. (FUENTE)
Organization: Foundation for the study of VTE diseases. (FUENTE) (Other)
Other Study IDs: PIv9042015
Record Dates: First submitted 2016-07-06; First posted 2016-07-14 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Computerized Registry of Patients with Venous Thromboembolism (RIETE) is a multidisciplinary Project initiated in march 2001 and consisting in obtaining an extensive data registry of consecutive patients with venous thromboembolism.

The main objective is to provide information on the Internet to help physicians to improve their knowledge on the natural history of thromboembolic disease, particularly in those subgroups of patients who are usually not recruited in randomized clinical trials (pregnant women, elderly patients, disseminated cancer, severe renal insufficiency, patients with contraindications to anticoagulation therapy, extreme body weight, etc), with the purpose of decreasing mortality, frequency of thromboembolic recurrences as well as bleeding complications and arterial events.

As an additional objective RIETE is also aimed to create predictive scores that help physicians to better identify patients with high risk of presenting some of these complications.

The primary parameters recorded by the registry comprise details of each patient's clinical status, including any coexisting or underlying conditions, and the type, dose, duration and outcome (during the first 3 months of therapy) of antithrombotic treatment. Study endpoints are clinically recognized (and objectively confirmed) recurrences of VTE, major and minor bleeding complications, and death.

DETAILED DESCRIPTION:
The RIETE Registry pretends the improvement of care of patients with thromboembolic disease. Very often the investigators pose serious doubts on how to manage a specific patient. Sometimes because it is a patient with thrombocytopenia, a pregnant woman, a patient with a recent cerebral bleeding or cerebral metastasis, a patient with gastroduodenal ulcer or hepatic cirrhosis. There is no clinical evidence about how the investigators should manage these patients and the investigators have to individualize its management. The bibliography available is not of much help. Only if the investigators have a database with a sufficient number of cases, they may be able to make evidence based decisions.

This database on the Internet will allow the investigators to consult and obtain an immediate response when taking care of a patient who needs an individualized management. After introducing the patient the investigators will automatically obtain the data of all patients with similar clinical profiles. And this will help the investigators to identify high-risk patients and thus facilitate them preventing possible future complications.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed VTE (acute deep-vein thrombosis, pulmonary embolism and/or superficial venous thrombosis) by objective tests.
* Informed consent to the participation in the study, according to the requirements of the ethics committee within each hospital.

Exclusion Criteria:

* Participation in a therapeutic clinical trial with an unknown drug.
* Inability to the 3 month follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Venous Thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2001-03; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
VTE events and complications | 3 years
  Study endpoints are clinically recognized (and objectively confirmed) recurrences of VTE, major and minor bleeding complications, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Monreal, Study Chair — Foundation for the study of VTE diseases. (FUENTE)
Locations (256):
- United States (6):
  - Yale University School of Medicine, New Haven, Connecticut
  - College of Medicine - Jacksonville University of Florida, Jacksonville, Florida
  - Evanston NorthShore University HealthSystem, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Northwell Health System, Manhasset, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Clínica San Camilo, Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires
  - Clínica Privada Pueyrredón, Mar del Plata, Buenos Aires
- Medical University of Vienna, Vienna, Vienna, Austria
- Hospital UZ Leuven, Leuven, Leuven, Belgium
- Brazil (4):
  - Hospital Jorge Valente, Salvador, Estado de Bahia
  - Hospital Glória d'Or, Rio de Janeiro, Rio de Janeiro
  - Hospital Cardio Pulmonar, Salvador, Salvador
  - Botucatu Medical School - São Paulo State University (UNESP), Botucatu, São Paulo
- China (2):
  - The Seven Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality
- Colombia (4):
  - Hospital Universitario San Vicente Fundación, Medellín, Antioquia
  - Hospital Universitario Fundación Santa Fé de Bogota, Bogotá, Bogota D.C.
  - Hospital Universitario Fundación Valle del Lili, Cali, Colombia
  - Hospital Universitario San José de Buga Fundación, Guadalajara de Buga, Valle del Cauca Department
- Czechia (3):
  - University Hospital Hradec Kralove, Hradec Králové, Hradec Králové
  - Hospital Pardubická Krasjská Nemocnice A.S., Pardubice, Pardubice
  - University Hospital Plzen, Pilsen, Plzen
- Ecuador (3):
  - Hospital Luis Vernaza, Guayaquil, Guayas
  - Hospital Clínica La Merced, Quito, Quito
  - Hospital SOLCA Núcleo de Quito, Quito, Quito
- Ain Shams University Specialized Hospital, Cairo, Cairo Governorate, Egypt
- France (19):
  - University Hospital Jean Minjoz, Besançon, Besançon
  - CHRU Brest, Brest, Brest
  - Clermont-Ferrand University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes, Colombes
  - CHU de Dijon Bourgogne, Dijon, Dijon
  - Hôpital Édouard Herriot, Lyon, Lyon
  - Médipôle Hôpital Mutualiste, Villeurbanne, Lyon
  - Hôpital de la Timone, Marseille, Marseille
  - Hôpital Saint Eloi, Montpellier, Montpellier
  - CHU Nantes, Nantes, Nantes
  - Hôpital Europeen Georges Pompidou, Paris, Paris
  - Hôpital Lariboisiere, Paris, Paris
  - Hôpital Paris Saint-Joseph, Paris, Paris
  - Hôpital Saint-Louis, Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Pierre-Bénite
  - Hospital Center of Avignon, Avignon, Provenza
  - Institut Sainte Catherine, Avignon, Provenza
  - Hôpital Nord - CHU St-Etienne, Saint-Etienne, Saint-Etienne
  - Hôpital de Rangueil, Toulouse, Toulouse
- Municipal Hospital of Dresden Friedrichstadt, Dresden, Dresden, Germany
- Hospital Papageorgiou, Thessaloniki, Saloniki, Greece
- Hospital Escuela Universitario, Tegucigalpa, Francisco Morazán Department, Honduras
- Iran (6):
  - Imam Reza Hospital, Tabriz, East Azerbaijan Province
  - Abu-Ali- Sina Organ Transplant Center (OCT), Shiraz, Fars
  - Chamran Cardiology Hospital, Isfahan, Isfahan
  - Masih-Daneshvari Hospital, Tehran, Tehran Province
  - Rajaie Cardiovascular Medical and Research Center, Tehran, Tehran Province
  - Tehran Heart Center, Tehran, Tehran Province
- Mater Misericordiae University Hospital, Dublin, Leinster, Ireland
- Israel (4):
  - Rambam Healthcare Campus, Haifa, Haifa District
  - Galilee Medical Center, Nahariya, Nahariya
  - Hematology Institute of ZIV Medical Center, Safed, Safed
  - Sheba Medical Center, Ramat Gan, Tel Hashomer
- Italy (29):
  - Ospedale SS. Filippo e Nicola, Avezzano, Aquila
  - ULSS 1 Dolomiti, Belluno, Belluno
  - Spedali Civili di Brescia, Brescia, Brescia
  - AORN San Giuseppe Moscati Avellino, Avellino, Campania
  - Ospedale Buon Consiglio Fatebenefratelli, Naples, Campania
  - Hospital of Marcianise, Marcianise, Caserta
  - Ospedale CastelFranco Veneto, Castelfranco, Castelfranco Veneto
  - Istituti Ospitalieri di Cremona, Cremona, Cremona
  - Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Foggia
  - Ospedale Galliera, Genoa, Genova
  - A.O.U Policlinico "G. Martino", Messina, Messina
  - IRCCS Istituto Auxologico Italiano, Milan, Milan
  - Istituto Clinico Humanitas IRCCS, Rozzano, Milan
  - Federico II University Hospital, Naples, Naples
  - Presidio Ospedaliero Santa Maria Delle Grazie, Pozzuoli, Naples
  - Azienda Ospedaliera Universitaria di Parma, Parma, Parma
  - Azienda U.S.L. Di Ravenna - O.C. Di Faenza, Ravenna, Ravenna
  - Hospital Rieti, Rieti, Rieti
  - Ospedale Infermi, Rimini, Rimini
  - "A. Gemelli " Hospital, Rome, Rome
  - Ospedale San Camillo, Rome, Rome
  - Ospedale St. John, Rome, Rome
  - AOU S. Giovanni di Dio e Ruggi d´Aragona, Salerno, Salerno
  - Ospedale Santa Chiara di Trento, Trento, Trento
  - Ospedale Santa Maria della Misericordia, Udine, Udine
  - Università dell´Insubria, Varese, Varese
  - University of Padua, Padua, Veneto
  - Ospedale SS. Giovanni e Paolo di Venezia, Venice, Venice
  - Azienda ULSS 7 Pedemontana Regione Veneto, Santorso, Vicenza
- Japan (9):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka Saiseikai Noe Hospital, Osaka, Osaka
  - Japanese Red Cross Wakayama Medical Center, Wakayama, Wakayama
- Pauls Stradins Clinical University Hospital, Riga, Rīga, Latvia
- Hospital Central Universitario de Chihuahua, Chihuahua City, Chihuahua, Mexico
- Ibn Sina Hospital, Rabat, Rabat, Morocco
- North Macedonia (2):
  - PHI University Clinic of Pulmology and Allergy Skopje, Skopje, Grad Skopje
  - University Cardiology Clinic, Skopje, Grad Skopje
- Portugal (6):
  - Centro Hospitalar do Médio Ave, Vila Nova de Famalicão, Famalicão
  - Hospital Pedro Hispano - Unidade Local de Saúde de Matosinhos, Senhora da Hora, Matosinhos
  - Hospital General de Santo Antonio Porto, Porto, Porto District
  - Unidade Local de Saúde Entre Douro e Vouga, Santa Maria da Feira, Santa María Da Feira
  - Hospital García de Orta, Almada, Setúbal District
  - Centro Hospitalar Gaia/Espinho, EPE, Vila Nova de Gaia, Vila Nova de Gaia
- Spain (137):
  - Hospital Universitario A Coruña, A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Comarcal de Barbanza, Ribeira, A Coruña
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Albacete, Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario de Vinalopó, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Hospital de Poniente, El Ejido, Almería
  - Hospital Universitario de Badajoz, Badajoz, Badajoz
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Clínica Rotger, Palma de Mallorca, Balearic Islands
  - Hospital Municipal de Badalona, Badalona, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sant Celoni, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona, Barcelona
  - Hospital Universitario Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Vall d'Hebrón, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Consorci Hospitalari de Mataró, Mataró, Barcelona
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Parc Sanitari Sant Joan de Deu, Sant Boi de Llobregat, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Sant Joan Despí-Moisés Broggi, Sant Joan Despí, Barcelona
  - Hospital Sant Camil, Sant Pere de Ribes, Barcelona
  - Fundació Hospital del L'Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - Hospital Universitario Mutua Terrassa, Terrassa, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Comarcal de L'Alt Penedés, Vilafranca del Penedès, Barcelona
  - Hospital Universitario de Burgos, Burgos, Burgos
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital General Universitari de Castelló, Castellon, Castellón
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Virgen de Altagracia, Manzanares, Ciudad Real
  - Hospital Santa Bárbara, Puertollano, Ciudad Real
  - Hospital General Virgen de la Luz, Cuenca, Cuenca
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Hospital Infanta Margarita, Cabra, Córdoba
  - Hospital de la Cruz Roja de Córdoba, Córdoba, Córdoba
  - Hospital San Juan de Dios, Córdoba, Córdoba
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital de Montilla, Montilla, Córdoba
  - Hospital de Figueres, Figueres, Gerona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Gerona
  - Hospital d'Olot i Comarcal de la Garrotxa, Olot, Gerona
  - Hospital de Palamós, Palamós, Gerona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitario de Guadalajara, Guadalajara, Guadalajara
  - Hospital Universitario de Donostia, San Sebastián, Guipúzcoa
  - Hospital de Zumarraga, Zumarraga, Guipúzcoa
  - Hospital de Can Misses, Ibiza Town, Ibiza
  - Hospital del Alto Guadalquivir Andújar, Jaén, Jaen
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Fundación Hospital Calahorra, Calahorra, La Rioja
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Doctor José Molina Orosa, Arrecife, Lanzarote
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Complejo Hospitalario Insular-Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Hospital del Tajo, Aranjuez, Madrid
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Monográfico ASEPEYO, Coslada, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - S&H Medical Science Service, Madrid, Madrid
  - Hospital Central de la Defensa Gómez Ulla, Madrid, Madrid
  - Hospital de Cantoblanco, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Vithas Madrid La Milagrosa, Madrid, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Comarcal de la Axarquía, Vélez-Málaga, Malaga
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Rafael Méndez de Lorca, Lorca, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital General Universitario Reina Sofía, Murcia, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Virgen del Castillo, Yecla, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Reina Sofía, Tudela, Navarre
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Hospital de Manacor, Manacor, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario San Agustín, Avilés, Principality of Asturias
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Valle del Nalón, Langreo, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital General de Segovia, Segovia, Segovia
  - Hospital Universitario de Valme, Seville, Sevilla
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital El Vendrell, El Vendrell, Tarragona
  - Hospital Univ. Joan XXIII de Tarragona, Tarragona, Tarragona
  - Pius Hospital de Valls, Tarragona, Tarragona
  - Hospital de Tortosa Verge de la Cinta, Tortosa, Tarragona
  - Hospital Comarcal de Alcañiz, Alcañiz, Teruel
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Lluis Alcanyis, Xàtiva, Valencia
  - Hospital Recoletas Campo Grande, Valladolid, Valladolid
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital Ernest Lluch Martin, Calatayud, Zaragoza
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital Universitario Araba, Vitoria-Gasteiz, Álava
- Switzerland (3):
  - University Hospital of Geneva, Geneva, Canton of Geneva
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Lausanne
- Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, Tyne Y Wear, United Kingdom
- Vietnam (5):
  - Bach Mai Hospital Vietnam Heart Institue, Hanoi, Hanoi
  - Hanoi Medical University Hospital, Hanoi, Hanoi
  - Huu Nghi Hospital, Hanoi, Hanoi
  - Viet Duc Hospital, Hanoi, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City, Ho Chi Minh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cohen O, Waldman Radinsky L, Kenet G, Mahe I, Barillari G, Soler S, Siguenza P, Del Valle Morales M, Villares P, Monreal M. Venous thromboembolism characteristics and outcomes among RIETE patients tested and untested for inherited thrombophilia. Blood Adv. 2024 Sep 24;8(18):4950-4959. doi: 10.1182/bloodadvances.2024012611. PMID 38669351
- [Derived] Bertoletti L, Madridano O, Jimenez D, Muriel A, Bikdeli B, Ay C, Trujillo-Santos J, Bosevski M, Siguenza P, Monreal M. Cancer-Associated Thrombosis: Trends in Clinical Features, Treatment, and Outcomes From 2001 to 2020. JACC CardioOncol. 2023 Nov 15;5(6):758-772. doi: 10.1016/j.jaccao.2023.09.003. eCollection 2023 Dec. PMID 38205016
- [Derived] Martin Romero M, Salazar Rosa V, Demelo Rodriguez P, Visona A, Farfan Sedano AI, Peris Sifre ML, Skride A, Usandizaga E, Meireles J, Monreal M. Clinical characteristics and outcomes in patients with retinal vein occlusion. Vasc Med. 2022 Dec;27(6):590-592. doi: 10.1177/1358863X221122505. Epub 2022 Sep 30. No abstract available. PMID 36178134
- [Derived] Prandoni P, Pesavento R, Bilora F, Fernandez Reyes JL, Madridano O, Soler S, Monreal M. No difference in outcome between therapeutic and preventive anticoagulation in patients with superficial vein thrombosis involving the saphenous-femoral junction. Vasc Med. 2022 Jun;27(3):290-292. doi: 10.1177/1358863X211066962. Epub 2022 Jan 30. No abstract available. PMID 35098818
- [Derived] Bikdeli B, Moustafa F, Nieto JA, Lee AI, Ruiz-Gimenez N, Lorenzo A, Schellong S, Soler S, Ortiz S, Morales MDV, Bosevski M, Gavin O, Lip GYH, Monreal M; RIETE Investigators. Clinical characteristics, time course, and outcomes of major bleeding according to bleeding site in patients with venous thromboembolism. Thromb Res. 2022 Mar;211:10-18. doi: 10.1016/j.thromres.2022.01.007. Epub 2022 Jan 14. PMID 35051831
- [Derived] Martinez-Urbistondo D, de la Garza RG, Villares-Fernandez P, Font C, Schellong S, Lopez-Nunez JJ, Gil-Diaz A, Del Carmen Diaz-Pedroche M, Hirmerova J, Monreal M; RIETE Investigators. Liver status and outcomes in patients without previous known liver disease receiving anticoagulant therapy for venous thromboembolism. Intern Emerg Med. 2022 Apr;17(3):725-734. doi: 10.1007/s11739-021-02858-x. Epub 2021 Oct 9. PMID 34626318
- [Derived] Exposito-Ruiz M, Arcelus JI, Caprini JA, Lopez-Espada C, Bura-Riviere A, Amado C, Loring M, Mastroiacovo D, Monreal M; RIETE Investigators. Timing and characteristics of venous thromboembolism after noncancer surgery. J Vasc Surg Venous Lymphat Disord. 2021 Jul;9(4):859-867.e2. doi: 10.1016/j.jvsv.2020.11.017. Epub 2020 Nov 26. PMID 33248295
- [Derived] Camporese G, Simioni P, Di Micco P, Fernandez-Capitan C, Rivas A, Font C, Sahuquillo JC, Villares P, Prandoni P, Monreal M; RIETE Investigators. Edoxaban for the Long-Term Therapy of Venous Thromboembolism: Should the Criteria for Dose Reduction be Revised? Clin Transl Sci. 2021 Jan;14(1):335-342. doi: 10.1111/cts.12876. Epub 2020 Oct 10. PMID 33038286
- [Derived] Jimenez D, Bikdeli B, Quezada A, Muriel A, Lobo JL, de Miguel-Diez J, Jara-Palomares L, Ruiz-Artacho P, Yusen RD, Monreal M; RIETE investigators. Hospital volume and outcomes for acute pulmonary embolism: multinational population based cohort study. BMJ. 2019 Jul 29;366:l4416. doi: 10.1136/bmj.l4416. PMID 31358508
- [Derived] Mellado M, Trujillo-Santos J, Bikdeli B, Jimenez D, Nunez MJ, Ellis M, Marchena PJ, Vela JR, Clara A, Moustafa F, Monreal M; RIETE Investigators. Vena cava filters in patients presenting with major bleeding during anticoagulation for venous thromboembolism. Intern Emerg Med. 2019 Oct;14(7):1101-1112. doi: 10.1007/s11739-019-02077-5. Epub 2019 May 3. PMID 31054013